CLINICAL TRIAL: NCT04124068
Title: Efficacy of GLO Science Professional Teeth Whitening Product Offerings in Adults
Brief Title: Efficacy of Teeth Whitening Product Offerings in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glo Science, Inc. (Industry)
Collaborators: Arizona School of Dentistry & Oral Health, A. T. Still University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLO-003
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Tooth Discoloration
Keywords: Teeth whitening; Teeth bleaching; Tooth discoloration
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (5):
- GLO Science Professional Chairside Teeth Whitening (Experimental)
  Interventions: Other: Hydrogen peroxide teeth whitening gel; Device: GLO Science Professional Teeth Whitening Device
- GLO Science Professional At-Home Teeth Whitening Device (Experimental)
  Interventions: Other: Hydrogen peroxide teeth whitening gel; Device: GLO Science Professional Teeth Whitening Device
- GLO Brilliant At-Home Teeth Whitening Device (Experimental)
  Interventions: Other: Hydrogen peroxide teeth whitening gel; Device: GLO Brilliant Teeth Whitening Device
- GLO Lit At-Home Teeth Whitening Device (Experimental)
  Interventions: Other: Hydrogen peroxide teeth whitening gel; Device: GLO Lit Teeth Whitening Device
- GLO Lit Whitening GLO Vials (Experimental)
  Interventions: Other: Hydrogen peroxide teeth whitening gel

INTERVENTIONS:
Other: Hydrogen peroxide teeth whitening gel — Hydrogen peroxide teeth whitening gel with concentrations ranging between 6% - 30%
Device: GLO Brilliant Teeth Whitening Device — Intra-oral mouthpiece connected to a battery in order to generate light and heat to effect the whitening treatment.
  Arms: GLO Brilliant At-Home Teeth Whitening Device
Device: GLO Lit Teeth Whitening Device — Intra-oral mouthpiece connected to a battery in order to generate light and heat to effect the whitening treatment.
  Arms: GLO Lit At-Home Teeth Whitening Device
Device: GLO Science Professional Teeth Whitening Device — Intra-oral mouthpiece connected to a battery in order to generate light and heat to effect the whitening treatment.
  Arms: GLO Science Professional At-Home Teeth Whitening Device; GLO Science Professional Chairside Teeth Whitening

SUMMARY:
This is a 30 day randomized, parallel comparative trial where participants with tooth shade of C2 or darker will be assigned to one of five groups. The participants will be evaluated for the difference in tooth shade, as determined by the digital VITA Easyshade V (provided by GLO) before the respective whitening regimen (baseline), immediately following the treatment period, and at 30 days (~4 weeks) from end of the treatment intervention.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate in the study.
* Be 18 to 65 years of age.
* Agree not to participate in any other oral/dental product studies during the trial.
* Agree to delay any elective dentistry (including dental prophylaxis) until the study has been completed.
* Agree to refrain from the use of any other teeth whitening products once assigned to a treatment group.
* Agree to refrain from the use of any oral care products that may cause staining (chlorhexidine rinses, stannous fluoride toothpaste, etc.).
* Agree to return for all scheduled visits and follow study procedures.
* Be in good general health, as determined by the investigator/designee based on a review of the health history/update for participation in the study.
* Have at least 4 gradable maxillary anterior teeth ( canine to canine) with a Vita Shade average score of C2 or darker.
* Be willing to refrain from consuming stain-causing food and beverages (i.e., coffee, tea, red wine, berries, etc.) during the initial treatment duration (treatment period excluding the 4 week follow up).
* Be a current or recent non-smoker (no smoking for at least 3 months).

Exclusion Criteria:

* Are undergoing treatment for gingivitis, periodontitis, or caries.
* Presence of self-reported tooth sensitivity.
* Present with fixed orthodontic appliances on the facial surfaces of the maxillary arch.
* Have dental crowns, veneers or composite restorations on gradable maxillary anterior teeth ( canine to canine) or mandibular anterior teeth.
* Have any oral pathologies or gross neglect of home care requiring prompt treatment, including periodontal disease, as evidenced by purulent exudate, exposed root surfaces (generalized recession), tooth mobility, and/or other signs indicating that the integrity of the data collected for that subject might be compromised.
* Present with any pre-existing oral or medical condition that the Investigator/designee determines may place the subject at increased health risk from study participation.
* Have meaningful malocclusion that would impact treatment or ease of viewing/scoring maxillary anterior teeth.
* Have teeth with severe or atypical intrinsic staining, such as that caused by tetracycline, fluorosis or hypocalcification.
* Have any known allergies to over-the-counter oral hygiene/whitening products.
* Have any known allergies to the trial product ingredients.
* Are pregnant and/or breastfeeding.
* Are current smokers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Tooth whitening efficacy: tooth shade value | Immediately following treatment period (32 minutes, 5 days or 7 days), and after 30 days
  Change in tooth shade value as indicated by the digital VITA Easyshade V

SECONDARY OUTCOMES:
Tooth whitening safety: presence/absence of adverse events | Immediately following treatment period (32 minutes, 5 days or 7 days), and after 30 days
  Post-treatment dentinal hypersensitivity and the presence/absence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ann Spolarich, RDH, PhD, Principal Investigator — Arizona School of Dentistry & Oral Health, A. T. Still University
Locations (1):
- Arizona School of Dentistry & Oral Health, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: No